CLINICAL TRIAL: NCT03019978
Title: Person-Centered Assessment and Monitoring Systems (PCAMS)
Brief Title: Person-Centered Assessment and Monitoring Systems
Acronym: PCAMS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Collaborators: Pennsylvania Bureau of Autism Services (Other)
Responsible Party: Principal Investigator, Michael Murray, Associate Professor of Psychiatry, Milton S. Hershey Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: STUDY00004326
Record Dates: First submitted 2017-01-11; First posted 2017-01-13 (Estimated); Last update posted 2020-04-08 (Actual); Status verified 2020-04

CONDITIONS: Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: PCAMS assessments — This is a longitudinal study, where data will be collected from 54 individuals who are already enrolled in Pennsylvania's ACAP program. Participants will be required to complete online assessments at baseline and then quarterly over a two-year time period.

SUMMARY:
The proposed study will include an analysis of data for residents of Pennsylvania who are age 21 and older, have a diagnosis of Autism Spectrum Disorder (ASD), and are enrolled in the Commonwealth's Adult Community Autism Program (ACAP). The individuals enrolled in the program will be administered a standardized assessment battery quarterly for two years. The proposed study will analyze the data gathered during each of the assessment periods in order to aid in service/treatment planning, assess for individual improvements, and ultimately measure treatment outcomes.

DETAILED DESCRIPTION:
The proposed study seeks to more closely monitor the changing needs and challenges of adults with ASD, which will be facilitated through a battery of assessments given over quarterly time points in a two year time period. Investigators seek to address whether increased frequency of behaviorally driven assessments will inform treatment. More specifically, investigators are interested in knowing if the assessment data influences treatment planning with providers or if it is guiding any decisions about treatment once data is returned to participants in a meaningful way which is easily understood. If data prompts treatment changes, the study will examine whether improvements are being shown months or even years later.

An "elected reporter", a family member, is asked to take part in the research study with the participant. An elected reporter is asked to complete several questionnaires quarterly, both reporting on themself and the participant.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled in Pennsylvania's Adult Community Autism Program (ACAP), > 18 years of age
* English as primary language spoken
* Ability to self-report (i.e. understand and answer assessment questions written at a third grade comprehension level)
* Have an Elected Reporter

Exclusion Criteria:

-Inability to provide consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-07; Primary Completion 2019-08 (Actual); Study Completion 2019-08 (Actual)

PRIMARY OUTCOMES:
Social Responsiveness Scale- 2 | annually over 2 years
Adult Behavior Checklist | annually over 2 years
Additional PROMIS measures | quarterly over 2 years
  Patient-Reported Outcomes Measurement Information System
Community Engagement measure | semi-annually over 2 years

SECONDARY OUTCOMES:
PROMIS measures | quarterly over 2 years
  Patient-Reported Outcomes Measurement Information System
Elected Reporter Community Engagement measure | semi-annually over 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Michael J Murray, M.D., Principal Investigator — Hershey Medical Center
Locations (1):
- The Penn State College of Medicine, Hershey, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No